CLINICAL TRIAL: NCT05970809
Title: A Randomised, Evaluator-Blinded, Two-Arm Study To Evaluate The Safety And Efficacy of a Novel Microneedle and Laser-Based Medical Device For The Treatment of Androgenetic Alopecia in Adult Males
Brief Title: Assessing the Safety and Efficacy of a Novel Microneedling and Laser Device for Male Pattern Hair Loss
Acronym: CS-SAGA-001
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: StimuSIL (Industry)
Collaborators: Ankara City Hospital Bilkent (Other); Istanbul University - Cerrahpasa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CS-SAGA-001
Record Dates: First submitted 2023-07-20; First posted 2023-08-01 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Male Pattern Baldness; Androgenetic Alopecia; Hair Loss/Baldness; Hair Loss; Pattern Baldness
Keywords: lasers; laser therapy; low-level light therapy; Low-Power Laser Therapy; Photobiomodulation Therapy; Low-Level Laser Therapy; Laser Biostimulation; LLLT; microtrauma, physical
MeSH Terms: conditions — Alopecia; Microtrauma, Physical

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants will be randomly allocated at a 1:1 ratio to receive treatment with Device type A or B.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Device A (Experimental): Device configuration A has metal and novel microneedles and lasers.
  Interventions: Device: SAGA-001 (A)
- Device B (Experimental): Device configuration B has novel microneedles and lasers.
  Interventions: Device: SAGA-001 (B)

INTERVENTIONS:
Device: SAGA-001 (A) — Use of a novel microneedle and laser device as a treatment for male patten hair loss with additional microwounding.
  Arms: Device A
Device: SAGA-001 (B) — Use of a novel microneedle and laser device as a treatment for male patten hair loss without additional microwounding.
  Arms: Device B

SUMMARY:
The purpose of this 24-week study is to see if the SAGA-001 device is safe and effective at helping people with male pattern hair loss.

Two different device configurations are being explored as part of this study. Device A has novel microneedles, lasers, and additional metal microneedles, while Device B only has novel microneedles and lasers.

Participants will receive 12 treatments with either Device A or Device B over the course of 24 weeks. Treatments will be performed on-site every two weeks.

DETAILED DESCRIPTION:
Participants will have the medical tests or procedures described below:

* Subjects will be asked about their previous medical history and current medications.
* Brief physical examinations will be performed, including a visual inspection of the scalp.
* Questions about medical history (including previous and current medication use) will be asked.
* Two types of photos will be taken: 1) "global photos", which are general photos of the subject's scalp, and 2) "macro photos", which are close-up photos of a part of the subject's scalp.
* Questions about treatment-related issues or unpleasantness will be asked.
* Subjects will be asked to rate the improvement they see in their photos.
* Subjects will be asked to rate their satisfaction with the treatment.

Participants will also be asked to record changes in medications, changes in medical treatments, and major life changes (such as major dietary changes, exercise changes, changes in life stressors, etc.) in a diary for the duration of treatment. They should also make note of any suspected side effects or issues they believe are related to the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing to sign an informed consent form
* Subject is within the age group of 22-55 years (including both ages)
* Subject is male
* Subject has AGA with a Stage IIa-V Hamilton-Norwood classification
* Subject's skin is within Fitzpatrick Skin Types I-IV

Exclusion Criteria:

* Subjects who have used any formulation or application/administration or type of treatment for disorders of the skin or scalp within 180 days prior to screening, including but not limited to the following treatments:

  1. Anti-inflammatory medications, including topical steroids
  2. Antifungal
  3. Skin, nail, hair rejuvenation supplementation, or IV infusions (includes vitamin, minerals, herbals, etc.)
  4. Hair growth shampoos, conditioners, and topicals
  5. Topical, dermal or oral minoxidil, finasteride, or dutasteride
  6. Hair growth stimulation treatments, i.e. PRP, stem cells, exosomes, growth factors, microneedling, mesotherapy
  7. LED or low level laser therapy treatments, ie. laser helmets, laser caps, and laser combs
  8. Infrared saunas
* Subjects with alopecia other than AGA, such as alopecia areata, alopecia totalis, telogen effluvium, anagen effluvium, and acquired cicatricial alopecia
* Subjects with a history of bleeding disorders
* Subjects on anticoagulant medications (aspirin, warfarin, heparin)
* Subject on autoimmune suppressant medications or suffering autoimmune diseases (e.g. humira)
* Subjects with an active infection at the local site
* Subjects with keloidal tendencies
* Subjects with chronic dermatological conditions affecting the scalp (e.g. eczema, psoriasis, etc.)
* Subjects with hepatic or renal disease, epilepsy, or any other major medical illness*
* Subjects that have undergone evaluation to rule out other causes of hair loss, because underlying causes (e.g., iron deficiency, lupus, thyroid disease, telogen effluvium, post-pregnancy, polycystic ovary, chemotherapy, etc.) would preclude assessment of performance in an androgenetic alopecia trial
* Subjects who are photosensitive or are using photosensitive drugs or topicals.
* Subjects who are taking anxiolytics medications
* Subjects who have been on hormone inhibitors or on hormone replacement therapy in the last 180 days
* Subjects who are at high risk of seizures
* Subjects who have a malignancy or a history of malignancies affecting the scalp
* Subjects that have undergone hair transplantation, scalp reduction, radiation to the scalp or chemotherapy within their lifetime.
* Subjects with current hair weaves, hair extensions, scalp tattoos, or who use occlusive wigs.
* Subjects who have used semi-permanent hair products (e.g. color, texturizers or relaxers) within 30 days prior to screening.
* Subjects with hair shorter than one-half inch (approximately 1.2 cm).
* Subjects who are unable to make regular follow-up visits.
* Subjects who are immediate family members (spouse, parent, child, or sibling; biological or legally adopted) of personnel directly affiliated with the study at the investigative sites, or individuals who are directly affiliated with the study at the investigative sites, or individuals directly affiliated with the study sponsor.

Ages: 22 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-10-24 (Actual)

PRIMARY OUTCOMES:
Change in terminal hair density | 24 weeks
  Changes in terminal hair density at the 24-week time point compared to baseline will be investigated using a binomial test for one proportion at a one-sided alpha with a 95% exact confidence interval, considering pi ≥ 60%, where pi is the true percentage of responders in the study population.
Change in terminal hair density | 16 weeks
  Changes in terminal hair density at the 16-week time point compared to baseline will be investigated using a binomial test for one proportion at a one-sided alpha with a 95% exact confidence interval, considering pi ≥ 60%, where pi is the true percentage of responders in the study population.

SECONDARY OUTCOMES:
Change in hair thickness | 16 weeks
  Increases and/or decreases in hair diameter at the 16-week time point compared to baseline will be investigated using a paired t-test at a one-sided alpha and a 95% confidence interval for mean change.
Change in hair thickness | 24 weeks
  Increases and/or decreases in hair diameter at the 24-week time point compared to baseline will be investigated using a paired t-test at a one-sided alpha and a 95% confidence interval for mean change.

CONTACTS AND LOCATIONS:
Overall Officials: Server Serdaroğlu, MD, Principal Investigator — İstanbul Üniversitesi Cerrahpaşa Tıp Fakültesi
Locations (2):
- Turkey (Türkiye) (2):
  - Ankara Bilkent Şehir Hastanesi Dermatoloji Klini, Ankara
  - İstanbul Üniversitesi Cerrahpaşa Tıp Fakültesi, Dahili Tıp Bilimleri Bölümü Deri ve Zührevi Hastalıklar Ana Bilim Dalı Kocamustafa Paşa, Istanbul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: StimuSIL's website — https://stimusil.com/